CLINICAL TRIAL: NCT07008586
Title: The Acute and Chronic Effects of OliPhenolia® Supplementation on Exercise Induced Inflammation and Functional Movement in Healthy Adult Humans.
Brief Title: The Impact of OliPhenolia® Supplementation on Exercise Induced Inflammation and Functional Movement in Humans.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Fattoria La Vialla di Gianni, Antonio e Bandino Lo Franco Soc. Agr. Sempl. (Unknown)
Responsible Party: Principal Investigator, Justin Roberts, Professor, Anglia Ruskin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ETH2425-3172
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Hydroxytyrosol; Exercise; Inflammation; Mobility
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Taste

STUDY DESIGN:
Intervention Model Description: Phase 1: Participants are randomly assigned OliPhenolia or placebo (matched in taste and appearance) in a double blind manner. Following a ≥7 day wash out period, participants then cross-over to the alternate product. Phase 2: Following a further ≥7 day wash out period, participants will continue to consume the same product (OliPhenolia or placebo) for a further 16 days ahead of final exercise assessments.
Who Masked: Participant, Investigator
Masking Description: Nutritional supplement is provided in a double-blind manner. Both participants and research testers will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OliPhenolia (Experimental): Commercially available concentrated olive fruit wastewater (OliPhenolia®) will be provided in a dose relative to participant body mass. In this arm, to assess the acute effects, participants will consume an oral bolus of 1.0mg∙kg-1 olive derived hydroxytyrosol via OliPhenolia® ahead of the exercise test. Following a wash out and necessary cross-over, participants will consume two doses of 1.0mg∙kg-1 olive derived hydroxytyrosol via OliPhenolia® daily for 16 days to assess the chronic component of this study..
  Interventions: Dietary Supplement: OliPhenolia®
- Placebo (Placebo Comparator): In this arm, to assess the acute component, participants will consume a single oral bolus of placebo (matched for taste and appearance to OliPhenolia®) ahead of the exercise test. The volume of this will be prepared by an independent researcher to match the specific volume of OliPhenolia® required for each participant. Following a wash out and necessary cross-over, participants will consume two doses placebo (identical volume to the acute component) daily for 16 days to assess the chronic component of this study.
  Interventions: Dietary Supplement: Taste and appearance matched placebo

INTERVENTIONS:
Dietary Supplement: OliPhenolia® — Olive derived hydroxytyrosol will be ingested via a commercially available olive fruit wastewater (OliPhenolia®) in a dose relative to participant body mass.
  Arms: OliPhenolia
Dietary Supplement: Taste and appearance matched placebo — Equal parts prune juice (Sunsweet California Prune Juice, Yuba City, CA, USA), diet cola (Tesco Cola, Tesco, UK) and tonic water (Tesco low calorie Indian tonic water, Tesco, UK).
  Arms: Placebo

SUMMARY:
This research proposal follows on from previously undertaken work investigating a commercially available olive derived product (OliPhenolia®) on potential exercise / functional benefits for healthy adults. Previous research investigated a dose response bioavailability of the main polyphenol in OliPhenolia® and related metabolites. Based on this data, the current study will aim to investigate, for the first time, whether the polyphenols in the product can positively influence exercise specific inflammation which may be pertinent to improving exercise recovery and is of current scientific interest. As such this research aims to understand the short term (Phase 1) and longer term (Phase 2) use of OliPhenolia® on acute recovery from a standard exercise bout.

Research questions:

1. Does an acute dose of OliPhenolia® reduce exercise associated inflammation markers and enhance functional recovery in healthy adult humans?
2. Does a consecutive 16 day intake of OliPhenolia® reduce exercise associated inflammation markers and enhance functional recovery in healthy adult humans?
3. Does a continued intake of OliPhenolia® during the recovery period after the exercise bout further amplify functional benefits compared experimental control?

Proposed methodology:

Phase 1 - To answer research question 1, following a randomisation procedure, participants will be allocated product (OliPhenolia®) or colour and taste matched placebo. A single serve of product (no more than 1.5 mg/kg of hydroxytyrosol (HT) via OliPhenolia®) or placebo will be provided ~40 minutes prior to a standardised exercise protocol. Resting wholeblood samples will be collected at 0 (baseline) +1, +24, +48 and +72 hours following the exercise bout to identify the impact of an acute dose of OliPhenolia® has on selected inflammatory biomarkers. This phase will be a placebo-controlled crossover design and therefore after a ≥7 day wash out period, participants will return to the exercise laboratory (Compass House Human Physiology laboratories, Anglia Ruskin University, Cambridge), supplement the alternate product and repeat the experimental protocol as outlined above.

Phase 2 - To answer research question 2, having completed Phase 1 (and following another ≥7 day wash out period), all participants will continue onto Phase 2, maintaining their previously assigned product, but this time will continue supplementation for 16 consecutive days. Phase 2 is therefore a parallel placebo-controlled design that focusses on a chronic supplementation of OliPhenolia®. Participants will consume one serve of either product or placebo twice daily for 16 days. After 16 days of supplementation participants will return to the exercise laboratory, and in the same manner as Phase 1, consume a single dose of their assigned product or placebo ~ 40 minutes prior to the standardised exercise protocol. Resting wholeblood samples will be collected following exercise at baseline, +1, +24, +48 and +72 hours.

To answer research question 3, all participants will be informed that they may be asked to consume an additional three days supplementation in a random manner (total 19 days). To limit participant burden 50 % of the experimental group (those that have been supplementing OliPhenolia®) and placebo group will continue supplementing two doses daily for the three days following the standardised exercise protocol (the three days where blood samples occur) in order to understand if a sustained course of OliPhenolia® can reduce the time taken for inflammatory mediators to return to baseline values.

DETAILED DESCRIPTION:
Following the current scientific interest surrounding the application of polyphenols in an exercise domain, the primary objectives of this research will build upon previously published work investigating polyphenol rich olive fruit water by identifying the acute and chronic effect of OliPhenolia® on inflammation and functional mobility following exercise induced inflammation. For the purpose of this research, the impact on inflammation will be investigated via the measurements of biomarkers Interleukin (IL)-6, IL-1ra, and Transforming growth factor-beta. Additionally, lactate dehydrogenase (a marker of muscle damage) and superoxide dismutase (a marker of oxidative stress) will also be measured to confirm the source and impact of the exercise induced inflammation. Furthermore, for the purpose of this research, a functional movement screen, localised goniometry and algometry will be measured surrounding the standardised exercise protocol to assess the impact of OliPhenolia on functional mobility. Within this study, participants will be required to attend a pre-screening and familiarisation session followed by three separate trials. Each trial, separated by a ~7 day wash out period will consist of four visits. The first visit (estimated duration 3 hours) will include the baseline resting venepuncture blood sample (0), basic physiological, anthropometric and cognitive assessments, standardised exercise protocol, post exercise blood sample (+1 hour) and post exercise physiological assessment. The standardised exercise protocol that will take place 40 minutes after the supplementation of OliPhenolia is as follows: A maximum of six sets of 25 drop jumps wearing a weighted vest (7.5% body mass) from a height of 60 cm with a maximum 10 second interval between jumps and a 1 min passive rest between sets (modified from Kirby et al., 2011). The following three visits (estimated duration 45 minutes) will take place over the following three days and require a resting venepuncture blood sample (+24 hours, +48 hours and +72 hours) and basic physiological assessment only. Prior to each visit, participants will be required to record a three-day habitual food and exercise diary and adhere to a prescribed low polyphenol meal the night before each laboratory visit. These measures are in place to increase the control of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 in line with manufacturer recommendations.
* Written informed consent.
* Willingness and ability to conform to the full protocol (please see full protocol).
* Judged by the investigator to be in good health.
* To have a pre-study health screen signed off by the lead researcher.

Exclusion Criteria:

* Current or recent (within the last 4 weeks) engagement with a strict dietary regime i.e., vegetarian / vegan / ketogenic / paleolithic / high protein / weight loss.
* Any known issues with blood taking.
* Any known bleeding disorders.
* Any known allergy to olives, grapes, lemon, coca cola or prunes.
* Average alcohol use of <21 glasses per week for men and <14 glasses per week for women (on average for the last six months).
* Any drug or medicine abuse in the last six months
* Known cardiovascular disease, disease related to the immune system (including HIV and hepatitis) and / or the respiratory system.
* Known Diabetes Mellitus type I or type II.
* Known renal or liver issues or known thyroid dysfunction.
* Currently undertaking regular heavy and / or extreme exercise (please discuss with the lead researcher if you are unsure).
* Current smoker or stopped smoking for <one month prior to the first visit.
* Current participation in any other clinical study within the month previous to the study start date (discuss with the lead researcher if unsure).
* Known pregnancy and / or lactation (women only)
* Uncertainty about the willingness or ability of the subject to comply with the protocol requirements.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Interleukin 6 | Four days
Interleukin 1 receptor antagonist | Four days
Transforming growth factor-beta | Four days
Lactate dehydrogenase | Four days
Superoxide dismutase | Four days

SECONDARY OUTCOMES:
Functional movement screen | Four days
  The functional movement screen (FMS) will utilise the FMS test kit (Functional Movement Systems s Inc, USA) and comprise of seven movement screens described by the creators of the method: (1) "Deep squat"; (2) "Hurdle step"; (3) "In-line lunge"; (4) "Shoulder mobility"; (5) "Active straight-leg raise"; (6) "Trunk stability push-up"; And (7) "Rotary stability. This test will be utilised to correlate to day-today functional movements through the assessment of hamstring and lumbar flexibility, whole body range of motion, core strength and stability.
Counter movement jump | Four days
  To assess lower body mechanical capacity and neuromuscular fatigue. Each participant will be invited to complete three repetitions of the counter movement jump with the highest repetition being recorded as the result.
Physical Readiness Questionnaire | Four days
  Participants will complete the European Federation of Sports Medicine Association (EFSMA) Pre-Participation Evaluation (PPE) form for recreationally active athletes (2021) to evaluate physical readiness. Section three of this form will be repeated to subjectively measure musculoskeletal soreness surrounding the standardised exercise bout. It is important to mention, this document is merely a guideline and the 'Medical' 'Laboratory tests' and 'Exercise Capacity' sections of this document within section 3 will not be used.
Perceived Muscle soreness | Four days
  Perceived muscle soreness of the lower body will be assessed using a visual analogue scale surrounding the standardised exercise protocol. Participants will subjectively rate their level of soreness during a maximal contraction of their quadriceps group by drawing an intersecting line across a continuum line extending from 0 cm (0 = no soreness) to 13 cm (13 = extreme soreness) (Buford et al. 2009). The scale is a continuous line and does not contain any segments or labels that would allow for quantification by the participant, therefore not allowing the participant to retain any perceived soreness value between testing sessions.
Pain questionnaire | Four days
  The McGill Pain Questionnaire will be employed to offer a subjective measure of musculoskeletal pain. The questionnaire that provides a list of 78 descriptors of pain from which the user can pick words that can later be summed to yield a sensory, effective, and evaluative overall pain score.
Algometry | Four days
  Participants perception of muscle soreness will be assessed using a simple handheld algometer (Wagner Instruments) in the non-dominant quadricep (thigh muscle). This device has been used numerous times within research studies in our laboratory. Data will be collected surrounding the standardised exercise protocol. Muscle soreness will be assessed using a standard process employing both pressure tolerance (reporting the maximum amount of pressure generating perceived discomfort that is tolerable) and secondly, pressure threshold (the minimum amount of force applied until the first verbal report of discomfort) is observed).
Range of motion at the knee and hip joint (Goiniometry) | Four days
  In order to obtain an objective measure of joint angle and range of motion in the hip and knee joint, a manual goniometer will be employed. Data will be collected at baseline, after the standardised exercise protocol as well as the three days following.
Cognitive Function | Four days
  The Mini Mental State Examination (MMSE), or similar, will be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Assessments of cognition will take place at baseline, 24, 48 and 72 hours following the standardised exercise protocol.
Heart Rate Variability | Four days
  Heart Rate Variability will be measured using a heart rate monitor to provide an objective physiological measure that is linked to the cardiovascular (CV) system and CV health.

CONTACTS AND LOCATIONS:
Overall Officials: Justin D Roberts, Professor, Principal Investigator — Anglia Ruskin University
Locations (1):
- Cambridge Centre for Sport and Exercise Sciences, Anglia Ruskin University,, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts JD, Lillis JB, Pinto JM, Chichger H, Lopez-Samanes A, Coso JD, Zacca R, Willmott AGB. The Effect of a Hydroxytyrosol-Rich, Olive-Derived Phytocomplex on Aerobic Exercise and Acute Recovery. Nutrients. 2023 Jan 13;15(2):421. doi: 10.3390/nu15020421. PMID 36678293